CLINICAL TRIAL: NCT07007832
Title: The Diagnostic Value of Bile-based Omics Analysis for Indeterminate Biliary Strictures
Brief Title: Bile Omics for Diagnosing Indeterminate Biliary Strictures
Status: Recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other); Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaobo Cai, Chief Physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: [2025] No. 236
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cholangiocarcinoma; Gallbladder Cancer and Extrahepatic Cholangiocarcinoma; Pancreatic Cancer; Bile Duct Strictures of Unknown Origin; Bile Duct Strictures
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms; Pancreatic Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde; Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- indeterminate biliary strictures: Pathologically or clinical confirmed
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiopancreatography — Since patients with biliary strictures almost universally require endoscopic biliary interventions for both diagnostic and drainage purposes, bile aspiration can be readily obtained during these procedures, facilitating subsequent analyses. However, proteomic and metabolomic profiling of bile in malignant biliary strictures remains unreported to date. This study aims to evaluate the diagnostic value of combining bile proteomics/metabolomics with biliary brush cytology/biopsy for malignant biliary strictures, while also providing evidence for identifying potential biomarkers.
  Other Names: biliary brush cytology; biopsy

SUMMARY:
The diagnosis of malignant biliary strictures remains a challenging aspect of biliary endoscopy. Molecular biological testing techniques based on bile have been reported to improve detection rates. However, whether the combination of bile-based omics studies and biliary brush cytology/biopsy can enhance diagnostic sensitivity has not yet been reported. This study aims to collect bile from patients with malignant biliary strictures, screen for molecular markers associated with biliary malignancies through multi-omics analysis, and subsequently validate these markers to establish a bile-based molecular diagnostic model.

ELIGIBILITY:
Inclusion Criteria:

* Indeterminate biliary strictures
* Aged 18-90 years
* Underwent ERCP with biliary biopsy and/or brush cytology

Exclusion Criteria:

* Coagulation disorders
* Pregnancy
* Malignancies of other organs unrelated to biliary strictures
* Declined participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in top-tier academic medical center in Shanghai, China (Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; The Third Affiliated Hospital of Naval Medical University; Shanghai Sixth People's Hospital, Shanghai Jiao Tong University School of Medicine)
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity | histologically or cytogically confirmed , or followed up for 6 months

SECONDARY OUTCOMES:
accuracy | histologically or cytologically confirmed or followed up for 6 months
Specificity | histologically or cytologically confirmed or followed up for 6 months
Positive predictive value, | histologically or cytologically confirmed or followed up for 6 months
negative predictive value | histologically or cytologically confirmed or followed up for 6 months
AUC area (histologically or cytologically confirmed or followed up for 6 months) | up for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xueying Ding, MD, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share de-identified IPD upon reasonable request after publication, contingent on approval from our institutional ethics committee. Data availability will be subject to a formal data use agreement to ensure patient confidentiality and compliance with local regulations. Restrictions may apply to protect participant privacy given the sensitive nature of clinical biliary data.

REFERENCES:
- [Background] Bhawal R, Oberg AL, Zhang S, Kohli M. Challenges and Opportunities in Clinical Applications of Blood-Based Proteomics in Cancer. Cancers (Basel). 2020 Aug 27;12(9):2428. doi: 10.3390/cancers12092428. PMID 32867043
- [Background] Arechederra M, Rullan M, Amat I, Oyon D, Zabalza L, Elizalde M, Latasa MU, Mercado MR, Ruiz-Clavijo D, Saldana C, Fernandez-Urien I, Carrascosa J, Jusue V, Guerrero-Setas D, Zazpe C, Gonzalez-Borja I, Sangro B, Herranz JM, Purroy A, Gil I, Nelson LJ, Vila JJ, Krawczyk M, Zieniewicz K, Patkowski W, Milkiewicz P, Cubero FJ, Alkorta-Aranburu G, G Fernandez-Barrena M, Urman JM, Berasain C, Avila MA. Next-generation sequencing of bile cell-free DNA for the early detection of patients with malignant biliary strictures. Gut. 2022 Jun;71(6):1141-1151. doi: 10.1136/gutjnl-2021-325178. Epub 2021 Jul 20. PMID 34285068
- [Background] Singhi AD, Nikiforova MN, Chennat J, Papachristou GI, Khalid A, Rabinovitz M, Das R, Sarkaria S, Ayasso MS, Wald AI, Monaco SE, Nalesnik M, Ohori NP, Geller D, Tsung A, Zureikat AH, Zeh H, Marsh JW, Hogg M, Lee K, Bartlett DL, Pingpank JF, Humar A, Bahary N, Dasyam AK, Brand R, Fasanella KE, McGrath K, Slivka A. Integrating next-generation sequencing to endoscopic retrograde cholangiopancreatography (ERCP)-obtained biliary specimens improves the detection and management of patients with malignant bile duct strictures. Gut. 2020 Jan;69(1):52-61. doi: 10.1136/gutjnl-2018-317817. Epub 2019 Apr 10. PMID 30971436
- [Background] de Oliveira PVAG, de Moura DTH, Ribeiro IB, Bazarbashi AN, Franzini TAP, Dos Santos MEL, Bernardo WM, de Moura EGH. Efficacy of digital single-operator cholangioscopy in the visual interpretation of indeterminate biliary strictures: a systematic review and meta-analysis. Surg Endosc. 2020 Aug;34(8):3321-3329. doi: 10.1007/s00464-020-07583-8. Epub 2020 Apr 27. PMID 32342216
- [Background] Platt KD, Schulman AR. Increasing the Yield: When More Is Better. Am J Gastroenterol. 2022 May 1;117(5):729-730. doi: 10.14309/ajg.0000000000001724. Epub 2022 Mar 14. PMID 35287142
- [Background] Wang J, Xia M, Jin Y, Zheng H, Shen Z, Dai W, Li X, Kang M, Wan R, Lu L, Hu B, Wan X, Cai X. More Endoscopy-Based Brushing Passes Improve the Detection of Malignant Biliary Strictures: A Multicenter Randomized Controlled Trial. Am J Gastroenterol. 2022 May 1;117(5):733-739. doi: 10.14309/ajg.0000000000001666. Epub 2022 Feb 2. PMID 35108222
- [Background] Korc P, Sherman S. ERCP tissue sampling. Gastrointest Endosc. 2016 Oct;84(4):557-71. doi: 10.1016/j.gie.2016.04.039. Epub 2016 May 6. No abstract available. PMID 27156656
- [Background] Elmunzer BJ, Maranki JL, Gomez V, Tavakkoli A, Sauer BG, Limketkai BN, Brennan EA, Attridge EM, Brigham TJ, Wang AY. ACG Clinical Guideline: Diagnosis and Management of Biliary Strictures. Am J Gastroenterol. 2023 Mar 1;118(3):405-426. doi: 10.14309/ajg.0000000000002190. Epub 2023 Jan 17. PMID 36863037
- [Background] Fujii-Lau LL, Thosani NC, Al-Haddad M, Acoba J, Wray CJ, Zvavanjanja R, Amateau SK, Buxbaum JL, Wani S, Calderwood AH, Chalhoub JM, Coelho-Prabhu N, Desai M, Elhanafi SE, Fishman DS, Forbes N, Jamil LH, Jue TL, Kohli DR, Kwon RS, Law JK, Lee JK, Machicado JD, Marya NB, Pawa S, Ruan W, Sawhney MS, Sheth SG, Storm A, Thiruvengadam NR, Qumseya BJ; (ASGE Standards of Practice Committee Chair [2020-2023]). American Society for Gastrointestinal Endoscopy guideline on role of endoscopy in the diagnosis of malignancy in biliary strictures of undetermined etiology: methodology and review of evidence. Gastrointest Endosc. 2023 Nov;98(5):694-712.e8. doi: 10.1016/j.gie.2023.06.007. Epub 2023 Jun 10. PMID 37307901
- See also: Diagnostic Efficacy of a Novel Rotating Brush for Endoscopic Sampling of Malignant Biliary Strictures: A Multicenter Prospective Study — https://journals.lww.com/ajg/abstract/2024/10000/diagnostic_efficacy_of_a_novel_rotating_brush_for.28.aspx
- See also: More Endoscopy-Based Brushing Passes Improve the Detection of Malignant Biliary Strictures: A Multicenter Randomized Controlled Trial — https://journals.lww.com/ajg/abstract/2022/05000/more_endoscopy_based_brushing_passes_improve_the.17.aspx